CLINICAL TRIAL: NCT02280447
Title: Safety and Immunogenicity of 3 Adjuvated Reduced Dose IPV-Al SSI Vaccines and Non-adjuvated Full Dose IPV SSI, Given as a Booster Vaccination to Adolescents With a History of IPV Vaccination at 3, 5, 12 Months and 5 Years of Age
Brief Title: 3 Adjuvated Reduced Dose IPV-Al SSI Vaccines and Non-adjuvated Full Dose IPV SSI, as Booster Vaccination to Adolescents
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Statens Serum Institut (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); CCBR Clinical Research (Unknown); Larix A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: VIPV-04; 2014-000052-29 (EudraCT Number)
Record Dates: First submitted 2014-10-29; First posted 2014-10-31 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Immunization, Booster

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1/3 IPV-Al SSI (Experimental): Reduced dose Al(OH)3 adjuvated IPV SSI with 1/3 of dose in full dose non-adjuvated IPV SSI (i.e.: Type 1:40 DU; Type 2:8 DU; Type 3:32 DU)
  1 X 0.5 mL suspension for injection for intramuscular use
  Interventions: Biological: 1/3 IPV-Al SSI, manufactured by SSI, Denmark
- 1/5 IPV-Al SSI (Experimental): Reduced dose Al(OH)3 adjuvated IPV SSI with 1/5 of dose in full dose non-adjuvated IPV SSI (i.e.: Type 1:40 DU; Type 2:8 DU; Type 3:32 DU)
  1 X 0.5 mL suspension for injection for intramuscular use
  Interventions: Biological: 1/5 IPV-Al SSI, manufactured by SSI, Denmark
- 1/10 IPV-Al SSI (Experimental): Reduced dose Al(OH)3 adjuvated IPV SSI with 1/10 of dose in full dose non-adjuvated IPV SSI (i.e.: Type 1:40 DU; Type 2:8 DU; Type 3:32 DU)
  1 X 0.5 mL suspension for injection for intramuscular use
  Interventions: Biological: 1/10 IPV-Al SSI, manufactured by SSI, Denmark
- IPV SSI (Active Comparator): Non-adjuvated full dose IPV SSI (i.e.: Type 1:40 DU; Type 2:8 DU; Type 3:32 DU)
  1 X 0.5 mL solution for injection for intramuscular use
  Interventions: Biological: IPV SSI, manufactured by SSI, Denmark

INTERVENTIONS:
Biological: 1/3 IPV-Al SSI, manufactured by SSI, Denmark — Intramuscular injection of 0.5 mL vaccine into deltoid muscle
  Other Names: Reduced dose (1/3) IPV adjuvated to Al(OH)3
  Arms: 1/3 IPV-Al SSI
Biological: 1/5 IPV-Al SSI, manufactured by SSI, Denmark — Intramuscular injection of 0.5 mL vaccine into deltoid muscle
  Other Names: Reduced dose (1/5) IPV adjuvated to Al(OH)3
  Arms: 1/5 IPV-Al SSI
Biological: 1/10 IPV-Al SSI, manufactured by SSI, Denmark — Intramuscular injection of 0.5 mL vaccine into deltoid muscle
  Other Names: Reduced dose (1/10) IPV adjuvated to Al(OH)3
  Arms: 1/10 IPV-Al SSI
Biological: IPV SSI, manufactured by SSI, Denmark — Intramuscular injection of 0.5 mL vaccine into deltoid muscle
  Other Names: Full dose inactivated polio vaccine, non-adjuvated
  Arms: IPV SSI

SUMMARY:
The background of the clinical trial is the overall aim of the World Health Organization (WHO) to obtain eradication of polio in the world. As part of this overall plan, inactivated polio vaccine (IPV) against poliovirus types 1, 2 and 3, at an affordable price, needs to become available in low resource third World countries.

The primary objective of the phase I/II clinical trial is to provide proof of concept (POC) that up to 10 times dose reduction of IPV SSI does not decrease the immunogenicity clinically significantly compared to full dose IPV SSI, by demonstrating the non-inferiority of the booster effects of each of 3 Al(OH)3 adjuvated reduced dose IPV formulations (1/3 IPV-Al SSI, 1/5 IPV-Al SSI and 1/10 IPV-Al SSI) compared to non-adjuvated full dose IPV SSI.

A total of 240 healthy adolescents with a history of IPV SSI vaccination at 3, 5, 12 months and 5 years of age according to the Danish vaccination program will be included in the trial.

DETAILED DESCRIPTION:
The trial is a phase I/II, parallel- and multi-group, randomised, controlled, multi-centre, non-inferiority trial investigating the safety and immunogenicity of 4 IPV vaccines, given as a booster vaccination to adolescents who have completed primary infant vaccination and pre-school booster vaccination with IPV in Denmark.

At Visit 1 (Screening and vaccination visit), written informed consent is obtained and the subject's eligibility is assessed according to the pre-specified in-/exclusion criteria, including measurement of oral temperature. If the subject is included, a pre-vaccination blood sample is taken for polio antibody determinations, and the subject is randomly allocated into one of the 4 groups to be vaccinated.

The subjects are observed for ½ an hour after the IMP injection and any immediate adverse events observed are to be recorded. A diary, thermometer and ruler are handed out to the subjects so that they can measure daily the injection site reactions and temperature the first 3 days (72 hours) and record any adverse event until the follow-up visit.

At Visit 2 (Follow-up visit), 28-35 days later, a post-vaccination blood sample is taken, the diary is collected, and adverse events and concomitant medications are recorded in the eCRF.

The trial is conducted in two parts. In the first part, 50 % of the subjects are randomised with allocation weights 4:4:1:1 to IPV SSI, 1/3 IPV-Al SSI, 1/5 IPV-Al SSI or 1/10 IPV-Al SSI, respectively. In the second part, the corresponding allocation weights are 1:1:4:4 for the remaining 50 % of the subjects.

After inclusion of 50 % of the subjects, an interim immunogenicity analysis is planned. While the interim analysis on 50% of the completed subjects is performed, the trial continues to recruit and randomise the remaining 50% of the subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Adolescents from ≥ 10 to ≤ 15 years of age at inclusion
2. Healthy assessed from medical history and oral temperature at inclusion
3. Vaccinated in Denmark according to the current vaccination program of 3 IPV doses in infancy and one IPV dose at pre-school age (i.e. born ≥ 1 July 1999)
4. Signed informed consent from adolescent's parent(s)/legal guardian(s)
5. Grant of authorised person's access to adolescent's medical records from adolescent's parent(s)/legal guardian(s)
6. Is willing and likely to comply with trial procedures

Exclusion Criteria:

1. Vaccinated with IPV ≤ 5 years prior to inclusion
2. Vaccinated with OPV any time prior to inclusion
3. Travelled in wild polio virus endemic region ≤ 5 years prior to inclusion
4. History of serious adverse reaction(s) after any previous vaccination
5. Known or suspected allergy to active or inactive vaccine constituents
6. Vaccinated with a live vaccine (e.g. measles, mumps, rubella, varicella, yellow fever or typhoid) ≤ 1 month prior to inclusion or during the trial. Subjects vaccinated with inactivated vaccines (e.g. tetanus, diphtheria, human papillomavirus, hepatitis A or B) are eligible for inclusion
7. Known or suspected immunodeficiency (e.g. HIV, leukaemia, lymphoma)
8. Severe uncontrolled disease (e.g. diabetes, asthma, epilepsy, heart or Crohn's disease). Patients in controlled medical treatment may be included, as assessed by the investigator
9. In treatment with systemic corticosteroids given p.o., i.v., i.m. ≤ 1 month prior to inclusion or during the trial. Subjects administered corticosteroid topically or by asthma inhalators are eligible for inclusion
10. In treatment with immune modulating products ≤ 3 months prior to inclusion or during the trial, e.g. blood products, immunoglobulins, cytostatics (e.g. methotrexate), TNF-antagonists (e.g. etanercerpt, infliximab, adalimumab, golimumab, certolizumab), or immunosuppressants (e.g. azathioprine or ciclosporin)
11. In treatment with any investigational medicinal product ≤ 3 months prior to inclusion or during the trial
12. A positive pregnancy test result at inclusion (for females who have had their first period) and/or objection to use contraception (for females who are sexually active)
13. Is unsuitable for participation in the trial or is not likely to comply with instructions as assessed by the investigator

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 240 (Actual)
Dates: Start 2014-11-13 (Actual); Primary Completion 2015-03 (Actual); Study Completion 2015-03-05 (Actual)

PRIMARY OUTCOMES:
Booster effect (day 28 / day 0 titres), from individual serum titre values for antibodies against poliovirus types 1, 2 and 3 measured in pre-vaccination and post-vaccination serum samples by a Vero Cell neutralising assay | On the day of and 28 days after the vaccination

SECONDARY OUTCOMES:
Seroconversion (≥ 4-fold day 28 / day 0 titre rise) rates, from individual serum titre values for antibodies against poliovirus types 1, 2 and 3 measured in pre-vaccination and post-vaccination serum samples by a Vero Cell neutralising assay | On the day of and 28 days after the vaccination
Frequencies of adverse events following the vaccination | On the day of and 28 days after the vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Line Markdanner Lindgren, Principal Investigator — Principal Investigator
Locations (3):
- Denmark (3):
  - CCBR, Aalborg
  - CCBR, Ballerup Municipality
  - CCBR, Vejle

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lindgren LM, Tingskov PN, Justesen AH, Nedergaard BS, Olsen KJ, Andreasen LV, Kromann I, Sorensen C, Dietrich J, Thierry-Carstensen B. First-in-human safety and immunogenicity investigations of three adjuvanted reduced dose inactivated poliovirus vaccines (IPV-Al SSI) compared to full dose IPV Vaccine SSI when given as a booster vaccination to adolescents with a history of IPV vaccination at 3, 5, 12months and 5years of age. Vaccine. 2017 Jan 23;35(4):596-604. doi: 10.1016/j.vaccine.2016.12.027. Epub 2016 Dec 24. PMID 28027810